CLINICAL TRIAL: NCT00167986
Title: Antibiotic Intervention Trial in a Medical Intensive Care Unit to Reduce the Acquisition of Vancomycin-Resistant Enterococci and ESBL Producing Escherichia Coli and Klebsiella Pneumoniae.
Brief Title: Study Evaluating Antibiotic Use in Reducing Vancomycin-Resistant Enterococci and ESBL Producing Escherichia Coli and Klebsiella Pneumoniae in Intensive Care
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 101498
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2007-03-15 (Estimated); Status verified 2007-03

CONDITIONS: Escherichia Coli Infections; Klebsiella Infections
Keywords: Bacterial Infections
MeSH Terms: conditions — Escherichia coli Infections; Klebsiella Infections; Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Drug: vancomycin-resistant enterococci and ESBL

SUMMARY:
To determine whether the restriction of 3rd generation cephalosporins and carbapenems contribute to the reduction of intestinal colonization or infection with vancomycin-resistant enterococci (VRE) in a medical intensive care unit (MICU).

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to or transferred to the MICU.
* Patients 18 years of age or older.
* Provide written informed consent.

Exclusion Criteria:

* Patients known to be infected or colonized by VRE or ESBL-producing E.coli, K.pneumoniae.
* Patients who have hypersensitivity to penicillin.
* Any underlying conditions or diseases that will be ultimately fatal within 48 hours.
* Any concurrent condition or medication which would interfere with absorption or metabolism of study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480
Dates: Start 2005-01

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Gyunggi-do, South Korea